CLINICAL TRIAL: NCT03841994
Title: Association of Gut Microbiome With Neonatal Complications and Neurodevelopment in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Professor, Seoul National University Hospital
Other Study IDs: 1801-128-917
Record Dates: First submitted 2019-02-01; First posted 2019-02-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Preterm Infants
Keywords: microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gastric juice, blood, stool, breast milk, transtracheal aspirates
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infant cohort: Preterm infants who were born <28 weeks of gestational age

SUMMARY:
A prospective cohort study investigating the effect of the formation of gut microbiome on the neonatal disease and the prognosis of neurodevelopment in preterm infants.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effect of the formation of gut microbiome on the neonatal disease and the prognosis of neurodevelopment in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants
* born less than 28+0 weeks gestation

Exclusion Criteria:

* Major congenital anomalies

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants who are born at < 28 weeks of gestation and admitted to the neonatal intensive care unit at Seoul national university children's hospital
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
The distribution rate of intestinal microbiome of stool by K-mer based taxonomic assignment | within 24 hours after birth
  Comparison of gut microbiome with 16s RNA gene specific sequencing in stool, breast milk, gastric juice
The distribution rate of intestinal microbiome of stool by K-mer based taxonomic assignment | 2 weeks after birth
  Comparison of gut microbiome with 16s RNA gene specific sequencing in stool, breast milk, gastric juice
The distribution rate of intestinal microbiome of stool by K-mer based taxonomic assignment | 3~5 weeks after birth
  Comparison of gut microbiome with 16s RNA gene specific sequencing in stool, breast milk, gastric juice
The distribution rate of intestinal microbiome of stool by K-mer based taxonomic assignment | at 37~40 weeks of postmenstrual age
  Comparison of gut microbiome with 16s RNA gene specific sequencing in stool, breast milk, gastric juice

SECONDARY OUTCOMES:
Brain MRI | at 37~40 weeks of postmenstrual age
  white matter injury
Bayley scales of infant and toddler development, third edition | at 18~24 months of corrected age
  For neurodevelopmental screening, Bayley scales of infant and toddler development, third edition yields composite scores for each cognitive, language, motor.
  It is considered normal when >85. Developmental delay is diagnosed when the mean result is below 85.
  Neurodevelopmental screening is considered normal when a child achieves these all.
Incidence of major morbidity | at 36~40 weeks of postmenstrual age
  Major morbidity such as bronchopulmonary dysplasia, periventricular leukomalacia, retinopathy of prematurity
Comparison of inflammation markers | with in 24 hours after birth, in 2 weeks, in 3~5 weeks, at 37~40 weeks of postmenstrual age
  Comparison of inflammation markers such as Interleukin(IL)-1 beta/IL-1F2, IL-6, IL-8/CXCL8, Tumor necrosis factor(TNF)-alpha, etc.
Comparison of short chain fatty acid at 4 period | with in 24 hours after birth, in 2 weeks, in 3~5 weeks, at 37~40 weeks of postmenstrual age
  Comparison of short chain fatty acid in stool and blood at 4 period

CONTACTS AND LOCATIONS:
Overall Officials: Ee-Kyung Kim, M.D., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao B, Stout MJ, Lee I, Mysorekar IU. Placental Microbiome and Its Role in Preterm Birth. Neoreviews. 2014 Dec 1;15(12):e537-e545. doi: 10.1542/neo.15-12-e537. PMID 25635174
- [Background] Choi Y, Kwon Y, Kim DK, Jeon J, Jang SC, Wang T, Ban M, Kim MH, Jeon SG, Kim MS, Choi CS, Jee YK, Gho YS, Ryu SH, Kim YK. Gut microbe-derived extracellular vesicles induce insulin resistance, thereby impairing glucose metabolism in skeletal muscle. Sci Rep. 2015 Oct 29;5:15878. doi: 10.1038/srep15878. PMID 26510393
- [Background] Cong X, Henderson WA, Graf J, McGrath JM. Early Life Experience and Gut Microbiome: The Brain-Gut-Microbiota Signaling System. Adv Neonatal Care. 2015 Oct;15(5):314-23; quiz E1-2. doi: 10.1097/ANC.0000000000000191. PMID 26240939
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] DiBartolomeo ME, Claud EC. The Developing Microbiome of the Preterm Infant. Clin Ther. 2016 Apr;38(4):733-9. doi: 10.1016/j.clinthera.2016.02.003. Epub 2016 Mar 2. PMID 26947798
- [Background] Kim MH, Rho M, Choi JP, Choi HI, Park HK, Song WJ, Min TK, Cho SH, Cho YJ, Kim YK, Yang S, Pyun BY. A Metagenomic Analysis Provides a Culture-Independent Pathogen Detection for Atopic Dermatitis. Allergy Asthma Immunol Res. 2017 Sep;9(5):453-461. doi: 10.4168/aair.2017.9.5.453. PMID 28677360
- [Background] Macfabe DF. Short-chain fatty acid fermentation products of the gut microbiome: implications in autism spectrum disorders. Microb Ecol Health Dis. 2012 Aug 24;23. doi: 10.3402/mehd.v23i0.19260. eCollection 2012. PMID 23990817
- [Background] Mshvildadze M, Neu J. The infant intestinal microbiome: friend or foe? Early Hum Dev. 2010 Jul;86 Suppl 1(Suppl 1):67-71. doi: 10.1016/j.earlhumdev.2010.01.018. Epub 2010 Feb 8. PMID 20116944
- [Background] Murgas Torrazza R, Neu J. The developing intestinal microbiome and its relationship to health and disease in the neonate. J Perinatol. 2011 Apr;31 Suppl 1:S29-34. doi: 10.1038/jp.2010.172. PMID 21448201
- [Background] Rea K, Dinan TG, Cryan JF. The microbiome: A key regulator of stress and neuroinflammation. Neurobiol Stress. 2016 Mar 4;4:23-33. doi: 10.1016/j.ynstr.2016.03.001. eCollection 2016 Oct. PMID 27981187
- [Background] Sanz Y. Gut microbiota and probiotics in maternal and infant health. Am J Clin Nutr. 2011 Dec;94(6 Suppl):2000S-2005S. doi: 10.3945/ajcn.110.001172. Epub 2011 May 4. PMID 21543533
- [Background] Stewart CJ, Embleton ND, Marrs EC, Smith DP, Nelson A, Abdulkadir B, Skeath T, Petrosino JF, Perry JD, Berrington JE, Cummings SP. Temporal bacterial and metabolic development of the preterm gut reveals specific signatures in health and disease. Microbiome. 2016 Dec 29;4(1):67. doi: 10.1186/s40168-016-0216-8. PMID 28034304
- [Background] Sung J, Kim N, Kim J, Jo HJ, Park JH, Nam RH, Seok YJ, Kim YR, Lee DH, Jung HC. Comparison of Gastric Microbiota Between Gastric Juice and Mucosa by Next Generation Sequencing Method. J Cancer Prev. 2016 Mar;21(1):60-5. doi: 10.15430/JCP.2016.21.1.60. Epub 2016 Mar 30. PMID 27051651
- [Background] Yoo JY, Rho M, You YA, Kwon EJ, Kim MH, Kym S, Jee YK, Kim YK, Kim YJ. 16S rRNA gene-based metagenomic analysis reveals differences in bacteria-derived extracellular vesicles in the urine of pregnant and non-pregnant women. Exp Mol Med. 2016 Feb 5;48(2):e208. doi: 10.1038/emm.2015.110. PMID 26846451
- [Background] Wang X, Buhimschi CS, Temoin S, Bhandari V, Han YW, Buhimschi IA. Comparative microbial analysis of paired amniotic fluid and cord blood from pregnancies complicated by preterm birth and early-onset neonatal sepsis. PLoS One. 2013;8(2):e56131. doi: 10.1371/journal.pone.0056131. Epub 2013 Feb 20. PMID 23437088
- [Result] Ardissone AN, de la Cruz DM, Davis-Richardson AG, Rechcigl KT, Li N, Drew JC, Murgas-Torrazza R, Sharma R, Hudak ML, Triplett EW, Neu J. Meconium microbiome analysis identifies bacteria correlated with premature birth. PLoS One. 2014 Mar 10;9(3):e90784. doi: 10.1371/journal.pone.0090784. eCollection 2014. PMID 24614698